CLINICAL TRIAL: NCT04034706
Title: Transcriptional and Epigenetic Program of PCOS Women
Acronym: EPIC
Status: Active, not recruiting | Type: Observational
Sponsor: AdventHealth Translational Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 1354588
Record Dates: First submitted 2019-07-24; First posted 2019-07-26 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: PCOS
MeSH Terms: interventions — Magnetic Resonance Spectroscopy; Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PCOS females: Females diagnosed with PCOS with a BMI between 23 and 40 kg/m2.
  Interventions: Other: DEXA; Other: Magnetic Resonance (MR) Assessment of the Abdomen; Other: MR assessment of Whole Body Fat; Procedure: Adipose tissue biopsy; Other: Oral glucose tolerance test
- Non-PCOS control females: Females without PCOS with a BMI between 23 and 40 kg/m2 split into 2 groups- apple shaped and pear shaped.
  Interventions: Other: DEXA; Other: Magnetic Resonance (MR) Assessment of the Abdomen; Other: MR assessment of Whole Body Fat; Procedure: Adipose tissue biopsy; Other: Oral glucose tolerance test

INTERVENTIONS:
Other: DEXA — DEXA Scans will be performed to measure body fat and estimate muscle mass using a General Electric Lunar iDXA whole-body scanner.
Other: Magnetic Resonance (MR) Assessment of the Abdomen — Include measures to assess liver lipid content and stiffness and perform volumetric fat quantitation.
Other: MR assessment of Whole Body Fat — Volumetric measurement of fat, muscle and bone
Procedure: Adipose tissue biopsy — 0.5 cm incision of the upper-outer right vastus lateralis, and either a 3-4mm Mercedes Liposuction needle, or a 4-6 mm Bergstrom needle will be inserted to aspirate approximately 7 grams of adipose tissue.
Other: Oral glucose tolerance test — Glucose tolerance will be assessed with a 75 g oral glucose tolerance test (OGTT). Subjects will be studied after an overnight fast.

SUMMARY:
The main goal is to reveal differences in global gene expression in two different adipose tissue (AT) depots of females with and without polycystic ovary syndrome (PCOS) and how these are influenced by upstream epigenetic markers

ELIGIBILITY:
Inclusion Criteria:

1. Women;
2. Age 18-45 years inclusive;
3. BMI 23-40 kg/m2 inclusive;
4. HbA1C ≤ 6.0% or fasting plasma glucose < 126 mg/dL;
5. Weight stable (± 3 kg) during the 3 months prior to enrollment;
6. Women must be > 9 months post-partum;
7. For PCOS: A documented history of PCOS from their physician according to the Androgen Excess (AE)-PCOS criteria: (defined by the presence of hyperandrogenism (clinical and/or biochemical), ovarian dysfunction (oligo-anovulation and/or polycystic ovaries), and the exclusion of related disorders (eg. hypoadrenalism, ovarian tumors)
8. Regular menstrual cycle for females without PCOS
9. Able to provide written, informed consent.

Exclusion Criteria:

1. Postmenopausal women
2. Women with hysterectomy
3. Pregnancy, lactation or < 9 months postpartum from the scheduled date of screening.
4. Fasting plasma glucose > 126 mg/dL, or HbA1c > 6% or diagnosis with Type 2 Diabetes (T2D) or Type 1 Diabetes (T1D)
5. History or presence of cardiovascular disease (unstable angina, myocardial infarction or coronary revascularization within 6 months, clinically significant abnormalities on EKG), presence of cardiac pacemaker, implanted cardiac defibrillator.
6. Liver disease (AST or ALT >2.5 times the upper limit of normal)
7. Kidney disease (creatinine >1.6 mg/dl or estimated GFR <60 ml/min)
8. Dyslipidemia, including triglycerides >500 mg/dl, LDL >200 mg/dl
9. Anemia (hemoglobin <11 g/dl)
10. Thyroid dysfunction (suppressed thyroid-stimulating hormone, elevated TSH <10 µIU/ml if symptomatic or elevated TSH >10 µIU/ml if asymptomatic)
11. Uncontrolled hypertension (BP >160 mmHg systolic or >100 mmHg diastolic)
12. Elevated hsCRP or known active infection
13. History of cancer within the last 5 years (skin cancers, with the exception of melanoma, may be acceptable)
14. History of drug or alcohol abuse (> 3 drinks per day) within the last 5 years. Current drug use may be determined by plasma or urine drug screens.
15. psychiatric disease prohibiting adherence to study protocol.
16. History of organ transplant.
17. Known history of HIV, active Hepatitis A, B or C or tuberculosis.
18. History of bariatric surgery.
19. Current smokers (smoking within the past 3 months).
20. Current use of beta-adrenergic blocking agents.
21. Use of oral or injectable anti-hyperglycemic agents: metformin, sulfonylureas, DPP IV inhibitors, SGLT-2 inhibitors, thiazolidinediones, acarbose, GLP-1 analogs and insulin unless willing to undertake a washout period of 15 days for metformin and GLP-1 analogs and undergo subsequent laboratory screening tests.
22. Gonadotropin Releasing Hormone (GnRH) and/or Antiandrogen use within the last 2 months.
23. Use of any medications known to influence fat and/or energy metabolism (eg growth hormone therapy, glucocorticoids [steroids], etc.)
24. Initiation or change in hormone replacement therapy within the past 3 months (including, but not limited to thyroid hormone, estrogen replacement therapy or In Vitro Fertilization therapy).
25. Current treatment with blood thinners or antiplatelet medications that cannot be safely stopped for biopsy and testing procedures.
26. Not able or willing to have DXA scans or are above the acceptable weight limit (450 lbs) of the DXA scanner.
27. Presence of any condition that, in the opinion of the Investigators, compromises participant safety or data integrity or the participant's ability to complete study visits.
28. Not able to participate in MRI assessments due to:

    1. Metal implants (pacemaker, non-removable body piercings, aneurysm clips) based on Investigator's judgment at screening
    2. Physical limitations or equipment tolerances (e.g., MRI bore size) based on Investigator's judgment at screening
    3. Inability to tolerate MRI imaging without sedation or claustrophobia

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Recruitment methods utilized may include, but will not be limited to, the following: recruitment from within the AdventHealth Translational Research Institute's patient population: electronic medical records and database searches (including third party recruitment vendors); advertising in multiple media such as print ads, flyers, brochures, posters; radio ads; television spots; and internet/social media advertising.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2020-01-31 (Actual); Primary Completion 2023-04-12 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Epigenomic and transcriptomic differences in abdominal vs gluteal subcutaneous adipose tissue between females with and without polycystic ovary syndrome | 6 months after the last participant will be enrolled
  Epigenetic profiles (DNA methylation) and gene expression (RNA-seq) will be performed on whole tissue abdominal fat and gluteofemoral fat biopsies in addition to cultured pre-adipocytes and adipocytes.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Smith, MD, Principal Investigator — Principal Investigator
Locations (1):
- AdventHealth Translational Research Institute, Orlando, Florida, United States

REFERENCES:
- [Background] Abbott DH, Barnett DK, Bruns CM, Dumesic DA. Androgen excess fetal programming of female reproduction: a developmental aetiology for polycystic ovary syndrome? Hum Reprod Update. 2005 Jul-Aug;11(4):357-74. doi: 10.1093/humupd/dmi013. PMID 15941725
- [Background] Abbott DH, Dumesic DA, Eisner JR, Colman RJ, Kemnitz JW. Insights into the development of polycystic ovary syndrome (PCOS) from studies of prenatally androgenized female rhesus monkeys. Trends Endocrinol Metab. 1998 Feb;9(2):62-7. doi: 10.1016/s1043-2760(98)00019-8. PMID 18406243
- [Background] Azziz R, Carmina E, Chen Z, Dunaif A, Laven JS, Legro RS, Lizneva D, Natterson-Horowtiz B, Teede HJ, Yildiz BO. Polycystic ovary syndrome. Nat Rev Dis Primers. 2016 Aug 11;2:16057. doi: 10.1038/nrdp.2016.57. PMID 27510637
- [Background] Barber TM, Golding SJ, Alvey C, Wass JA, Karpe F, Franks S, McCarthy MI. Global adiposity rather than abnormal regional fat distribution characterizes women with polycystic ovary syndrome. J Clin Endocrinol Metab. 2008 Mar;93(3):999-1004. doi: 10.1210/jc.2007-2117. Epub 2007 Dec 18. PMID 18089693
- [Background] Bjorntorp P. Adipose tissue distribution and function. Int J Obes. 1991 Sep;15 Suppl 2:67-81. PMID 1794941
- [Background] Bos G, Snijder MB, Nijpels G, Dekker JM, Stehouwer CD, Bouter LM, Heine RJ, Jansen H. Opposite contributions of trunk and leg fat mass with plasma lipase activities: the Hoorn study. Obes Res. 2005 Oct;13(10):1817-23. doi: 10.1038/oby.2005.221. PMID 16286530
- [Background] Ciaraldi TP, Aroda V, Mudaliar S, Chang RJ, Henry RR. Polycystic ovary syndrome is associated with tissue-specific differences in insulin resistance. J Clin Endocrinol Metab. 2009 Jan;94(1):157-63. doi: 10.1210/jc.2008-1492. Epub 2008 Oct 14. PMID 18854391
- [Background] de Koning L, Merchant AT, Pogue J, Anand SS. Waist circumference and waist-to-hip ratio as predictors of cardiovascular events: meta-regression analysis of prospective studies. Eur Heart J. 2007 Apr;28(7):850-6. doi: 10.1093/eurheartj/ehm026. Epub 2007 Apr 2. PMID 17403720
- [Background] Diamanti-Kandarakis E, Dunaif A. Insulin resistance and the polycystic ovary syndrome revisited: an update on mechanisms and implications. Endocr Rev. 2012 Dec;33(6):981-1030. doi: 10.1210/er.2011-1034. Epub 2012 Oct 12. PMID 23065822
- [Background] Divoux A, Karastergiou K, Xie H, Guo W, Perera RJ, Fried SK, Smith SR. Identification of a novel lncRNA in gluteal adipose tissue and evidence for its positive effect on preadipocyte differentiation. Obesity (Silver Spring). 2014 Aug;22(8):1781-5. doi: 10.1002/oby.20793. Epub 2014 May 23. PMID 24862299
- [Background] Elbers JM, Asscheman H, Seidell JC, Gooren LJ. Effects of sex steroid hormones on regional fat depots as assessed by magnetic resonance imaging in transsexuals. Am J Physiol. 1999 Feb;276(2):E317-25. doi: 10.1152/ajpendo.1999.276.2.E317. PMID 9950792
- [Background] Elbers JM, Asscheman H, Seidell JC, Megens JA, Gooren LJ. Long-term testosterone administration increases visceral fat in female to male transsexuals. J Clin Endocrinol Metab. 1997 Jul;82(7):2044-7. doi: 10.1210/jcem.82.7.4078. PMID 9215270
- [Background] Frayn KN. Adipose tissue as a buffer for daily lipid flux. Diabetologia. 2002 Sep;45(9):1201-10. doi: 10.1007/s00125-002-0873-y. Epub 2002 Jul 24. PMID 12242452
- [Background] Guo Z, Johnson CM, Jensen MD. Regional lipolytic responses to isoproterenol in women. Am J Physiol. 1997 Jul;273(1 Pt 1):E108-12. doi: 10.1152/ajpendo.1997.273.1.E108. PMID 9252486
- [Background] Horowitz JF, Klein S. Whole body and abdominal lipolytic sensitivity to epinephrine is suppressed in upper body obese women. Am J Physiol Endocrinol Metab. 2000 Jun;278(6):E1144-52. doi: 10.1152/ajpendo.2000.278.6.E1144. PMID 10827018
- [Background] Jason J. Polycystic ovary syndrome in the United States: clinical visit rates, characteristics, and associated health care costs. Arch Intern Med. 2011 Jul 11;171(13):1209-11. doi: 10.1001/archinternmed.2011.288. No abstract available. PMID 21747019
- [Background] Karastergiou K, Fried SK, Xie H, Lee MJ, Divoux A, Rosencrantz MA, Chang RJ, Smith SR. Distinct developmental signatures of human abdominal and gluteal subcutaneous adipose tissue depots. J Clin Endocrinol Metab. 2013 Jan;98(1):362-71. doi: 10.1210/jc.2012-2953. Epub 2012 Nov 12. PMID 23150689
- [Background] Kirchengast S, Huber J. Body composition characteristics and body fat distribution in lean women with polycystic ovary syndrome. Hum Reprod. 2001 Jun;16(6):1255-60. doi: 10.1093/humrep/16.6.1255. PMID 11387301
- [Background] Kokosar M, Benrick A, Perfilyev A, Fornes R, Nilsson E, Maliqueo M, Behre CJ, Sazonova A, Ohlsson C, Ling C, Stener-Victorin E. Epigenetic and Transcriptional Alterations in Human Adipose Tissue of Polycystic Ovary Syndrome. Sci Rep. 2016 Mar 15;6:22883. doi: 10.1038/srep22883. PMID 26975253
- [Background] Lavebratt C, Almgren M, Ekstrom TJ. Epigenetic regulation in obesity. Int J Obes (Lond). 2012 Jun;36(6):757-65. doi: 10.1038/ijo.2011.178. Epub 2011 Sep 13. PMID 21912396
- [Background] Manneras-Holm L, Leonhardt H, Kullberg J, Jennische E, Oden A, Holm G, Hellstrom M, Lonn L, Olivecrona G, Stener-Victorin E, Lonn M. Adipose tissue has aberrant morphology and function in PCOS: enlarged adipocytes and low serum adiponectin, but not circulating sex steroids, are strongly associated with insulin resistance. J Clin Endocrinol Metab. 2011 Feb;96(2):E304-11. doi: 10.1210/jc.2010-1290. Epub 2010 Nov 17. PMID 21084397
- [Background] Manolopoulos KN, Karpe F, Frayn KN. Gluteofemoral body fat as a determinant of metabolic health. Int J Obes (Lond). 2010 Jun;34(6):949-59. doi: 10.1038/ijo.2009.286. Epub 2010 Jan 12. PMID 20065965
- [Derived] Whytock KL, Divoux A, Sun Y, Hopf M, Yeo RX, Pino MF, Yu G, Smith SR, Walsh MJ, Sparks LM. Isolation of nuclei from frozen human subcutaneous adipose tissue for full-length single-nuclei transcriptional profiling. STAR Protoc. 2023 Mar 17;4(1):102054. doi: 10.1016/j.xpro.2023.102054. Epub 2023 Jan 20. PMID 36853719
- See also: Website for AdventHealth Translational Research Institute — https://www.adventhealth.com/research/translational-research-institute-metabolism-and-diabetes